CLINICAL TRIAL: NCT00353262
Title: An Open-label Study to Assess the Pharmacokinetic Interaction Between Xeloda and Oxaliplatin in Patients With Metastatic Colorectal Cancer.
Brief Title: A Study of Xeloda (Capecitabine) in Combination With Oxaliplatin in Patients With Metastatic Colorectal Cancer.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP18587
Record Dates: First submitted 2006-07-17; First posted 2006-07-18 (Estimated); Results first posted 2016-01-08 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Oxaliplatin; Capecitabine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Avastin; Drug: Oxaliplatin; Drug: capecitabine [Xeloda]

INTERVENTIONS:
Drug: Avastin — 7.5mg/kg iv (cycle 3 only)
Drug: Oxaliplatin — 130mg/m2 iv (cycles 1, 2 and 3)
Drug: capecitabine [Xeloda] — 1000mg/m2 po bid (cycles 1, 2 and 3)

SUMMARY:
This single arm study will investigate possible pharmacokinetic interactions between Xeloda and oxaliplatin, and assess whether the pharmacokinetics of Xeloda and/or oxaliplatin is influenced by the addition of Avastin. All subjects will provide samples for pharmacokinetic analysis during the first 3 cycles of treatment. In cycles 1 and 2 patients will receive a treatment regimen containing Xeloda (1000mg/m2 bid) and oxaliplatin (130mg/m2 iv) and in cycle 3 Avastin (7.5mg/kg iv) will be added to the regimen. The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* adenocarcinoma of colon or rectum, with metastatic or locally advanced disease.

Exclusion Criteria:

* previous systemic treatment for advanced or metastatic disease;
* previous treatment with oxaliplatin or Avastin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-07; Primary Completion 2006-09 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Canada (3):
  - Hamilton, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 36 participants were enrolled in this study at three sites in Canada between 8 August 2005 and 24 April 2008.
Groups:
- Capecitabine+ Oxaliplatin+ Bevacizumab: In Cycle 1, participants received a single oral dose of capecitabine 1000 milligrams per meter square (mg/m^2 on Day 1 followed by 2-hour intravenous (IV) infusion of oxaliplatin 130 mg/m^2 on Day 2 followed by oral dosing of capecitabine 1000 mg/m^2 twice-daily (BID) from Day 5 to Day 14 . In Cycle 2, participants received IV infusion of oxaliplatin 130 mg//m^2 over 2 hours on Day 1 along with capecitabine 1000 mg/m^2 orally BID until Day 14. In Cycle 3, participants received IV infusion of bevacizumab 7.5 mg/kg over 90 minutes on Day 1 at the same time as oxaliplatin 130 mg//m^2 was administered as an IV infusion over 2 hours (Day 1 every 3 weeks) along with capecitabine1000 mg//m^2 orally BID until Day 14. Treatment with the Cycle 3 dosing regimen continued for a further 13 cycles (i.e. Cycle 16) or until progressive disease or unacceptable toxicity or until the participant withdrew consent
Period: Overall Study
Arm/Group | Capecitabine+ Oxaliplatin+ Bevacizumab
Started | 36
Completed | 7
Not Completed | 29
Not completed — Adverse Event | 8
Not completed — Withdrawal by Subject | 2
Not completed — Insufficient Therapeutic Response | 13
Not completed — Progression | 1
Not completed — Surgery | 4
Not completed — Break from Chemotherapy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Capecitabine+ Oxaliplatin+ Bevacizumab
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.3 (13.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Area Under The Plasma Concentration-Time Curve From Zero To Infinity (AUC0-Inf) of 5'-Deoxy-5-fluorouridine 5'-(DFUR)
Description: AUC0-infinity represents the area under the concentration-time curve of the analyte (5'-DFUR) in plasma over the time interval from 0 extrapolated to infinity. The analyte 5'-DFUR, the direct precursor of 5-fluorouracil (5-FU), is considered to be the most important metabolite of capecitabine in plasma. The unit of measure was nanograms per millilitre per hour (ng/mL * hr).
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours post the dose.
Population: All patients for whom observations contributing to the relevant assessments were available, who did not experience dose reductions, and for whom dosing was as required by the protocol were included in the corresponding analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL*hr
Arm/Group | Capecitabine+ Oxaliplatin+ Bevacizumab
Number analyzed (Participants) | 26
ng/mL*hr
  Cycle 1, Day 1 | 13605 (33)
  Cycle 2, Day 1 | 12177 (27)
  Cycle 3, Day 1 | 11817 (38)
Statistical Analysis 1: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; Cycle 2, Day 1 versus Cycle 1, Day 1; Test type: Superiority or Other; Geometric mean ratio = 0.90, 90% CI 2-sided [0.79 to 1.02]
Statistical Analysis 2: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; Cycle 3, Day 1 versus Cycle 1, Day 1; Test type: Superiority or Other; Geometric mean ratio = 0.87, 90% CI 2-sided [0.76 to 0.99]
Statistical Analysis 3: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; Cycle 3, Day 1 to Cycle 2, Day 1; Test type: Superiority or Other; Geometric mean ratio = 0.97, 90% CI 2-sided [0.85 to 1.10]

2. Primary Outcome: AUC0-inf for Free Platinum
Description: AUC0-infinity represents the area under the concentration-time curve of the analyte (free platinum) in plasma over the time interval from 0 extrapolated to infinity. AUC0-inf for free platinum was calculated for each participant from the concentration-data obtained on Days 2 to 5 of Cycle 1, and Days 1 to 4 for Cycle 2 and 3. Free platinum is not bound to plasma proteins and is considered to be the most clinically significant measure of pharmacological and toxicological activity.
Time Frame: Predose , 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 and 72 hours from the beginning of the 2 hour oxaliplatin infusion on Days 2 to 5 of Cycle 1, and Days 1 to 4 for Cycle 2 and 3.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL * hr
Arm/Group | Capecitabine+ Oxaliplatin+ Bevacizumab
Number analyzed (Participants) | 26
ng/mL * hr
  Cycle 1, Day 2 | 10069 (23)
  Cycle 2 , Day 1 | 10537 (24)
  Cycle 3, Day 1. | 10225 (23)
Statistical Analysis 1: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; Cycle 2, Day 1 versus Cycle 1, Day 2; Test type: Superiority or Other; Geometric mean ratio = 1.05, 90% CI 2-sided [1.01 to 1.08]
Statistical Analysis 2: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; Cycle 3, Day 1 to Cycle 1, Day 2; Test type: Superiority or Other; Geometric mean ratio = 1.02, 90% CI 2-sided [0.98 to 1.05]
Statistical Analysis 3: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; Cycle 3, Day 1 to Cycle 2, Day 1; Test type: Superiority or Other; Geometric mean ratio = 0.97, 90% CI 2-sided [0.94 to 1.00]

3. Secondary Outcome: AUC (0-infinity) of Capecitabine and Its Metabolites (5'-DFCR, 5-FU, and FBAL)
Description: AUC0-infinity represents the area under the concentration-time curve of the analytes (5'-DFCR, 5-FU, and FBAL) in plasma over the time interval from 0 extrapolated to infinity. After oral administration, capecitabine is first metabolized in the liver to 5'-deoxy-5-fluorocytidine (5'-DFCR), which is then converted to 5'-DFUR, and then catalytically activated to 5-FU.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours post the dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL*hr
Arm/Group | Capecitabine+ Oxaliplatin+ Bevacizumab
Number analyzed (Participants) | 26
ng/mL*hr
  Capcetabine , Cycle 1, Day 1 | 5217 (57)
  Capcetabine , Cycle 2, Day 1 | 5299 (54)
  Capcetabine , Cycle 3, Day 1 | 6130 (68)
  5'-DFCR , Cycle 1, Day 1 | 7630 (76)
  5'-DFCR , Cycle 2, Day 1 | 6409 (47)
  5'-DFCR, Cylce 3, Day 1 | 7989 (52)
  5-FU , Cycle 1, Day 1 | 437 (92)
  5-FU , Cycle 2, Day 1 | 355 (50)
  5-FU , Cycle 3, Day 1 | 343 (86)
  FBAL , Cycle 1, Day 1 | 17904 (27)
  FBAL , Cycle 2, Day 1 | 17413 (26)
  FBAL , Cycle 3, Day 1 | 17356 (34)
Statistical Analysis 1: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; Capecitabine: Cycle 2, Day 1 versus Cycle 1, Day 1; Test type: Superiority or Other; Geometric mean ratio = 1.02, 90% CI 2-sided [0.83 to 1.24]
Statistical Analysis 2: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; Capecitabine: Cycle 3, Day 1 to Cycle 2, Day 1; Test type: Superiority or Other; Geometric mean ratio = 1.16, 90% CI 2-sided [0.94 to 1.42]
Statistical Analysis 3: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; Capecitabine: Cycle 3, Day 1 to Cycle 1, Day 1; Test type: Superiority or Other; Geometric mean ratio = 1.17, 90% CI 2-sided [0.96 to 1.44]
Statistical Analysis 4: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; 5'-DFCR: Cycle 2, Day 1 versus Cycle 1, Day 1; Test type: Superiority or Other; Geometric mean ratio = 0.86, 90% CI 2-sided [0.69 to 1.08]
Statistical Analysis 5: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; 5'-DFCR: Cycle 3, Day 1 versus Cycle 1, Day 1; Test type: Superiority or Other; Geometric mean ratio = 1.08, 90% CI 2-sided [0.86 to 1.34]
Statistical Analysis 6: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; 5'-DFCR: Cycle 3, Day 1 versus Cycle 2, Day 1; Test type: Superiority or Other; Geometric mean ratio = 1.25, 90% CI 2-sided [1.00 to 1.55]
Statistical Analysis 7: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; 5-FU: Cycle 2, Day 1 versus Cycle 1, Day 1; Test type: Superiority or Other; Geometric mean ratio = 0.81, 90% CI 2-sided [0.66 to 1.01]
Statistical Analysis 8: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; 5-FU: Cycle 3, Day 1 versus Cycle 1, Day 1; Test type: Superiority or Other; Geometric mean ratio = 0.79, 90% CI 2-sided [0.64 to 0.97]
Statistical Analysis 9: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; 5-FU: Cycle 3, Day 1 versus Cycle 2, Day 1; Test type: Superiority or Other; Geometric mean ratio = 0.97, 90% CI 2-sided [0.78 to 1.19]
Statistical Analysis 10: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; FBAL: Cycle 2, Day 1 versus Cycle 1, Day 1; Test type: Superiority or Other; Geometric mean ratio = 0.97, 90% CI 2-sided [0.91 to 1.04]
Statistical Analysis 11: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; FBAL: Cycle 3, Day 1 versus Cycle 1, Day 1; Test type: Superiority or Other; Geometric mean ratio = 0.97, 90% CI 2-sided [0.90 to 1.04]
Statistical Analysis 12: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; FBAL: Cycle 3, Day 1 versus Cycle 2, Day 1; Test type: Superiority or Other; Geometric mean ratio = 1.00, 90% CI 2-sided [0.93 to 1.07]

4. Secondary Outcome: AUC0-last of Capecitabine and Its Metabolites (5'-DFUR, 5'-DFCR, 5 FU, and FBAL)
Description: Area under the plasma concentration-time curve from time zero to the time of the last measurable plasma concentration time point of capecitabine and its metabolites (5'-DFUR, 5'-DFCR, 5 FU, and FBAL).
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours post the dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL*hr
Arm/Group | Capecitabine+ Oxaliplatin+ Bevacizumab
Number analyzed (Participants) | 26
ng/mL*hr
  5' DFUR , Cycle 1, Day 1 | 13503 (33)
  5' DFUR, Cycle 2 , Day 1 | 12057 (28)
  5' DFUR, Cycle 3, Day 1 | 11618 (38)
  Capecitabine, Cycle 1, Day 1 | 5201 (57)
  Capecitabine, Cycle 2, Day 1 | 5273 (54)
  Capecitabine, Cycle 3, Day 1 | 6093 (68)
  5'-DFCR, Cycle 1, Day 1 | 6150 (80)
  5'-DFCR, Cycle 2 , Day 1 | 6378 (47)
  5'-DFCR, Cycle 3, Day 1 | 7909 (52)
  5-FU, Cycle 1, Day 1 | 433 (92)
  5-FU, Cycle 2, Day 1 | 350 (51)
  5-FU, Cycle 3, Day 1 | 336 (84)
  FBAL, Cycle 1, Day 1 | 16773 (26)
  FBAL, Cycle 2, Day 1 | 15992 (26)
  FBAL, Cycle 3, Day 1 | 14947 (31)

5. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Capecitabine and Its Metabolites (5'-DFUR, 5'-DFCR, 5 FU, and FBAL)
Description: Cmax is defined as maximum observed analyte concentration of capecitabine and its metabolites (5'-DFUR, 5'-DFCR, 5 FU, and FBAL)
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours post the dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Capecitabine+ Oxaliplatin+ Bevacizumab
Number analyzed (Participants) | 26
ng/mL
  5'-DFUR, Cycle 1, Day 1 | 8847 (48)
  5'-DFUR , Cycle 2, Day 1 | 6545 (48)
  5'-DFUR , Cycle 3, Day 1 | 5693 (54)
  Capecitabine, Cycle 1, Day 1 | 4930 (72)
  Capecitabine, Cycle 2, Day 1 | 4065 (73)
  Capecitabine, Cycle 3, Day 1 | 4167 (81)
  5' DFCR, Cycle 1, Day 1 | 3902 (78)
  5' DFCR, Cycle 2, Day 1 | 3407 (66)
  5' DFCR , Cycle 3, Day 1 | 3747 (69)
  5-FU, Cycle 1 , Day 1 | 292 (63)
  5-FU, Cycle 2, Day 1 | 216 (63)
  5-FU, Cycle 3, Day 1 | 168 (83)
  FBAL, Cycle 1, Day 1 | 3970 (19)
  FBAL, Cycle 2, Day 1 | 3627 (27)
  FBAL, Cycle 3, Day 1 | 3292 (34)
Statistical Analysis 1: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; 5'-DFUR: Cycle 2, Day 1 versus Cycle 1, Day 1; Test type: Superiority or Other; Geometric mean ratio = 0.74, 90% CI 2-sided [0.61 to 0.90]
Statistical Analysis 2: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; 5'-DFUR: Cycle 3, Day 1 versus Cycle 1, Day 1; Test type: Superiority or Other; Geometric mean ratio = 0.64, 90% CI 2-sided [0.53 to 0.79]
Statistical Analysis 3: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; 5'-DFUR: Cycle 3, Day 1 versus Cycle 2, Day 1; Test type: Superiority or Other; Geometric mean ratio = 0.87, 90% CI 2-sided [0.71 to 1.06]
Statistical Analysis 4: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; Capecitabine: Cycle 2, Day 1 versus Cycle 1, Day 1; Test type: Superiority or Other; Geometric mean ratio = 0.82, 90% CI 2-sided [0.63 to 1.08]
Statistical Analysis 5: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; Capecitabine: Cycle 3, Day 1 versus Cycle 2, Day 1; Test type: Superiority or Other; Geometric mean ratio = 1.03, 90% CI 2-sided [0.78 to 1.34]
Statistical Analysis 6: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; Capecitabine: Cycle 3, Day 1 versus Cycle 1, Day 1; Test type: Superiority or Other; Geometric mean ratio = 0.85, 90% CI 2-sided [0.65 to 1.10]
Statistical Analysis 7: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; 5'-DFCR: Cycle 2, Day 1 versus Cycle 1, Day 1; Test type: Superiority or Other; Geometric mean ratio = 0.87, 90% CI 2-sided [0.65 to 1.18]
Statistical Analysis 8: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; 5'-DFCR: Cycle 3, Day 1 versus Cycle 1, Day 1; Test type: Superiority or Other; Geometric mean ratio = 0.96, 90% CI 2-sided [0.71 to 1.30]
Statistical Analysis 9: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; 5'-DFCR: Cycle 3, Day 1 versus Cycle 2, Day 1; Test type: Superiority or Other; Geometric mean ratio = 1.10, 90% CI 2-sided [0.81 to 1.49]
Statistical Analysis 10: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; 5-FU: Cycle 2, Day 1 versus Cycle 1, Day 1; Test type: Superiority or Other; Geometric mean ratio = 0.74, 90% CI 2-sided [0.56 to 0.98]
Statistical Analysis 11: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; 5-FU: Cycle 3, Day 1 versus Cycle 1, Day 1; Test type: Superiority or Other; Geometric mean ratio = 0.58, 90% CI 2-sided [0.44 to 0.76]
Statistical Analysis 12: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; 5-FU: Cycle 3, Day 1 versus Cycle 2, Day 1; Test type: Superiority or Other; Geometric mean ratio = 0.78, 90% CI 2-sided [0.59 to 1.03]
Statistical Analysis 13: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; FBAL: Cycle 2, Day 1 versus Cycle 1, Day 1; Test type: Superiority or Other; Geometric mean ratio = 0.91, 90% CI 2-sided [0.83 to 1.00]
Statistical Analysis 14: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; FBAL: Cycle 3, Day 1 versus Cycle 1, Day 1; Test type: Superiority or Other; Geometric mean ratio = 0.83, 90% CI 2-sided [0.76 to 0.91]
Statistical Analysis 15: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; FBAL: Cycle 3, Day 1 versus Cycle 2, Day 1; Test type: Superiority or Other; Geometric mean ratio = 0.91, 90% CI 2-sided [0.83 to 1.00]

6. Secondary Outcome: Elimination Half-life Period (t1/2 Beta) of Capecitabine and Its Metabolites (5'-DFUR , 5'-DFCR, 5 FU, and FBAL)
Description: t1/2 Beta is the time measured for the plasma concentration to decrease by 1 half to its original concentration of capecitabine and its metabolites (5'-DFUR , 5'-DFCR, 5 FU, and FBAL)
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours post the dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Capecitabine+ Oxaliplatin+ Bevacizumab
Number analyzed (Participants) | 26
hour
  5' DFUR; Cycle 1, Day 1 | 0.65 (19)
  5' DFUR, Cycle 2 , Day 1 | 0.64 (49)
  5' DFUR, Cycle 3, Day 1 | 0.75 (39)
  Capecitabine, Cycle 1, Day 1 | 0.37 (52)
  Capecitabine, Cycle 2, Day 1 | 0.51 (55)
  Capecitabine, Cycle 3, Day 1 | 0.56 (42)
  5'-DFCR, Cycle 1, Day 1 | 0.71 (33)
  5'-DFCR, Cycle 2 , Day 1 | 0.75 (32)
  5'-DFCR, Cycle 3, Day 1 | 0.79 (24)
  5-FU, Cycle 1, Day 1 | 0.61 (20)
  5-FU, Cycle 2, Day 1 | 0.67 (61)
  5-FU, Cycle 3, Day 1 | 0.71 (31)
  FBAL, Cycle 1, Day 1 | 2.77 (19)
  FBAL, Cycle 2, Day 1 | 2.68 (26)
  FBAL, Cycle 3, Day 1 | 2.64 (33)

7. Secondary Outcome: AUC0-infinity for Total Platinum
Description: AUC0-infinity represents the area under the concentration-time curve of the analyte (total platinum) in plasma over the time interval from 0 extrapolated to infinity.
Time Frame: Pre-dose, and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 and 72 hours from the beginning of the two hour oxaliplatin infusion on Days 2 to 5 of Cycle 1, and Days 1 to 4 for Cycle 2 and 3
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL* hr
Arm/Group | Capecitabine+ Oxaliplatin+ Bevacizumab
Number analyzed (Participants) | 26
ng/mL* hr
  Cycle 1, Day 2 | 139329 (24)
  Cycle 2, Day 1 | 167610 (17)
  Cycle 3, Day 1 | 186268 (21)
Statistical Analysis 1: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; Total Platinum: Cycle 2, Day 1 versus Cycle 1, Day 2; Test type: Superiority or Other; Geometric mean ratio = 1.20, 90% CI 2-sided [1.09 to 1.33]
Statistical Analysis 2: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; Total Platinum: Cycle 3, Day 1 versus Cycle 1, Day 2; Test type: Superiority or Other; Geometric mean ratio = 1.34, 90% CI 2-sided [1.21 to 1.48]
Statistical Analysis 3: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; Total Platinum: Cycle 3, Day 1 versus Cycle 2, Day 1; Test type: Superiority or Other; Geometric mean ratio = 1.11, 90% CI 2-sided [1.01 to 1.23]

8. Secondary Outcome: AUC0-last of Total And Free Platinum
Description: Area under the plasma concentration-time curve from time zero to the time of the last measurable plasma concentration time point of Total And Free Platinum.
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL* hr
Arm/Group | Capecitabine+ Oxaliplatin+ Bevacizumab
Number analyzed (Participants) | 26
ng/mL* hr
  Total Platinum: Cycle 1, Day 2 | 85406 (20)
  Total Platinum: Cycle 2, Day 1 | 97083 (12)
  Total Platinum: Cycle 3, Day 1 | 97011 (17)
  Free Platinum: Cycle 1, Day 2 | 9399 (24)
  Free Platinum: Cycle 2, Day 1 | 9818 (25)
  Free Platinum: Cycle 3, Day 1 | 9604 (22)

9. Secondary Outcome: Cmax of Total And Free Platinum
Description: Cmax is defined as maximum observed analyte concentration of Total And Free Platinum.
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Capecitabine+ Oxaliplatin+ Bevacizumab
Number analyzed (Participants) | 26
ng/mL
  Total Platinum: Cycle 1, Day 2 | 3652 (14)
  Total Platinum: Cycle 2, Day 1 | 3741 (19)
  Total Platinum: Cycle 3, Day 1 | 3706 (21)
  Free Platinum: Cycle 1, Day 2 | 1818 (27)
  Free Platinum: Cycle 2, Day 1 | 1840 (36)
  Free Platinum: Cycle 3, Day 1 | 1813 (30)
Statistical Analysis 1: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; Total Platinum: Cycle 2, Day 1 versus Cycle 1, Day 2; Test type: Superiority or Other; Geometric mean ratio = 1.02, 90% CI 2-sided [0.96 to 1.09]
Statistical Analysis 2: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; Total Platinum: Cycle 3, Day 1 versus Cycle 1, Day 2; Test type: Superiority or Other; Geometric mean ratio = 1.01, 90% CI 2-sided [0.95 to 1.08]
Statistical Analysis 3: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; Total Platinum: Cycle 3, Day 1 versus Cycle 2, Day 1; Test type: Superiority or Other; Geometric mean ratio = 0.99, 90% CI 2-sided [0.93 to 1.05]
Statistical Analysis 4: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; Free Platinum: Cycle 2, Day 1 versus Cycle 1, Day 2; Test type: Superiority or Other; Geometric mean ratio = 1.01, 90% CI 2-sided [0.94 to 1.09]
Statistical Analysis 5: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; Free Platinum: Cycle 3, Day 1 versus Cycle 1, Day 2; Test type: Superiority or Other; Geometric mean ratio = 1.00, 90% CI 2-sided [0.92 to 1.08]
Statistical Analysis 6: Comparison: Capecitabine+ Oxaliplatin+ Bevacizumab; Free Platinum: Cycle 3, Day 1 versus Cycle 2, Day 1; Test type: Superiority or Other; Geometric mean ratio = 0.99, 90% CI 2-sided [0.91 to 1.07]

10. Secondary Outcome: T1/2 Beta of Total And Free Platinum
Description: T1/2 beta is the time measured for the plasma concentration to decrease by 1 half to its original concentration of total and free platinum.
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Capecitabine+ Oxaliplatin+ Bevacizumab
Number analyzed (Participants) | 26
hour
  Total Platinum: Cycle 1, Day 2 | 48.70 (30)
  Total Platinum: Cycle 2, Day 1 | 55.73 (24)
  Total Platinum: Cycle 3, Day 1 | 67.28 (26)
  Free Platinum: Cycle 1, Day 2 | 17.64 (10)
  Free Platinum: Cycle 2, Day 1 | 18.41 (9)
  Free Platinum: Cycle 3, Day 1 | 18.47 (10.90)

11. Secondary Outcome: Volume of Distribution at Steady State (VSS) of Total And Free Platinum
Description: VSS is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state.
Time Frame: Pre-dose, and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48 and 72 hours
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | Capecitabine+ Oxaliplatin+ Bevacizumab
Number analyzed (Participants) | 26
mL
  Total Platinum: Cycle 1, Day 2 | 109007 (23)
  Total Platinum: Cycle 2, Day 1 | 105097 (21)
  Total Platinum: Cycle 3, Day 1 | 112141 (21)
  Free Platinum: Cycle 1, Day 2 | 387158 (23)
  Free Platinum: Cycle 2, Day 1 | 389193 (29)
  Free Platinum: Cycle 3, Day 1 | 401040 (24)

12. Secondary Outcome: Clearance of Total And Free Platinum
Description: CL is a calculation of the rate at which a drug is removed from the body via renal, hepatic and other clearance pathways, expressed as volume (milliliters) per unit of time (hour).
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/Hr
Arm/Group | Capecitabine+ Oxaliplatin+ Bevacizumab
Number analyzed (Participants) | 26
mL/Hr
  Total Platinum: Cycle 1, Day 2 | 1603 (78)
  Total Platinum: Cycle 2, Day 1 | 1331 (22)
  Total Platinum: Cycle 3, Day 1 | 1198 (25)
  Free Platinum: Cycle 1, Day 2 | 22183 (23)
  Free Platinum: Cycle 2, Day 1 | 21176 (26)
  Free Platinum: Cycle 3, Day 1 | 21823 (23)

13. Secondary Outcome: Number Of Participants With Adverse Events (AEs)
Description: An adverse event is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product. This includes any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Pre-existing conditions which worsened during the study were also to be reported as AEs.
Time Frame: Approximately 3 Years (up to 28 days after the last intake of study medication)
Population: All 36 participants who received at least one dose of capecitabine.
Measure: Number; unit: Participants
Arm/Group | Capecitabine+ Oxaliplatin+ Bevacizumab
Number analyzed (Participants) | 36
Participants
  Any AE | 36
  Any SAE | 16

14. Secondary Outcome: Marked Laboratory Abnormalities
Description: Number of participants with marked laboratory abnormalities (hematology, coagulation, liver function, renal function, protein, electrolytes, miscellaneous).
Time Frame: Up to 28 days after last chemotherapy administration
Population: All 36 participants who received at least one dose of capecitabine.
Measure: Number; unit: Participants
Arm/Group | Capecitabine+ Oxaliplatin+ Bevacizumab
Number analyzed (Participants) | 36
Participants
  Hematocrit - high | 2
  Hematocrit - low | 5
  Hemoglobin - low | 6
  Platelets - high | 1
  Platelets - low | 9
  RBC - low | 12
  WBC - high | 1
  WBC - low | 7
  Neutrophils - high | 1
  Neutrophils - low | 3
  PT (INR) - high | 2
  ASAT (SGOT) - high | 6
  LDH - high | 2
  ALAT (SGPT) - high | 7
  Alk. Phos. - high | 6
  Dir. Bilirubin - high | 3
  Total Bilirubin - high | 2
  Creatinine - high | 0
  Albumin - low | 4
  Potassium - low | 2
  Sodium - low | 2
  Calcium - low | 1
  Glucose Fasting - high | 4

ADVERSE EVENTS:
Time Frame: Approximately 3 Years (up to 28 days after the last intake of study medication)
Description: Adverse event is defined as any untoward medical occurrence in a patient or clinical investigation patient administered a pharmaceutical product and includes any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Arm/Group | Capecitabine+ Oxaliplatin+ Bevacizumab
Serious Adverse Events (participants affected / at risk) | 16/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine+ Oxaliplatin+ Bevacizumab (N=36)
Diarrhoea (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Enteritis (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 6
Pyrexia (General disorders) | 3
Pain (General disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine+ Oxaliplatin+ Bevacizumab (N=36)
Nausea (Gastrointestinal disorders) | 30
Diarrhoea (Gastrointestinal disorders) | 29
Vomiting (Gastrointestinal disorders) | 21
Abdominal pain (Gastrointestinal disorders) | 14
Constipation (Gastrointestinal disorders) | 10
Abdominal discomfort (Gastrointestinal disorders) | 7
Flatulence (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 5
Rectal haemorrhage (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 3
Haematochezia (Gastrointestinal disorders) | 3
Toothache (Gastrointestinal disorders) | 3
Anorectal discomfort (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Gastrooesophageal reflux Disease (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 2
Rectal Discharge (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 32
Temperature intolerance (General disorders) | 10
Mucosal inflammation (General disorders) | 9
Oedema peripheral (General disorders) | 7
Pyrexia (General disorders) | 4
Catheter site erythema (General disorders) | 3
Chills (General disorders) | 3
Injection site pain (General disorders) | 3
Pain (General disorders) | 3
Catheter related complication (General disorders) | 2
Catheter site rash (General disorders) | 2
Chest discomfort (General disorders) | 2
Injection site discolouration (General disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 22
Neuropathy peripheral (Nervous system disorders) | 14
Headache (Nervous system disorders) | 9
Paraesthesia (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 4
Ataxia (Nervous system disorders) | 2
Neuralgia (Nervous system disorders) | 2
Palmar-plantar (Skin and subcutaneous tissue disorders) | 20
Erythrodysaesthesia syndrome Dry skin (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 5
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 5
Nail disorder (Skin and subcutaneous tissue disorders) | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Joint stiffness (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Trismus (Musculoskeletal and connective tissue disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 20
Hypokalaemia (Metabolism and nutrition disorders) | 10
Dehydration (Metabolism and nutrition disorders) | 7
Hyponatraemia (Metabolism and nutrition disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Anxiety (Psychiatric disorders) | 7
Insomnia (Psychiatric disorders) | 7
Confusional state (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 3
Restlessness (Psychiatric disorders) | 2
Thrombosis (Vascular disorders) | 6
Hypertension (Vascular disorders) | 5
Flushing (Vascular disorders) | 3
Hypotension (Vascular disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 11
Anaemia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Lacrimation increased (Eye disorders) | 6
Vision blurred (Eye disorders) | 3
Gamma-glutamyltransferase increased (Investigations) | 2
Weight decreased (Investigations) | 2
Dysuria (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 2
Palpitations (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 2
Hypersensitivity (Immune system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.